CLINICAL TRIAL: NCT02965989
Title: Effectiveness of a Online Training Program With a Clinical Procedure Standardized: "Blood Culture in Units of Nursing". Quasi-experimental Study
Brief Title: Effectiveness of a Online Training Program With a Clinical Procedure Standardized in Units of Nursing (CPSUN)
Acronym: CPSUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ignacio Zaragoza García (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor-Investigator, Ignacio Zaragoza García, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: InveCuidSkill16
Record Dates: First submitted 2016-10-26; First posted 2016-11-17 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Infection Control; Preventive Measures
Keywords: nursery care; nursery infection; online learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online training of a nursing technique (Experimental): Participants receives an individual online training of extraction of blood culture for 3 months (This platform aims to improve knowledge and skills), they are sent 3 homework (one per month) and are evaluated at the end of each.
  Interventions: Procedure: Online training of a nursing technique
- not receive online training (No Intervention): Participants don´t receives an individual online training of extraction of blood culture.Do their work as usual.

INTERVENTIONS:
Procedure: Online training of a nursing technique — The professionals with participant in the experimental arm receive an online training of a technique of extraction of blood culture and other arm the professionals no receive any training. They work as usual.
  Other Names: Elsevier Clinical Skills
  Arms: Online training of a nursing technique

SUMMARY:
This study evaluates if the implementation of an online platform with procedures and protocols, improve the knowledge of professionals and can have a health impact related to decreased contamination of blood cultures.

DETAILED DESCRIPTION:
This is a Quasi-experimental study, with parallel groups (experimental and control).

The aim of this study is to evaluate the efficacy of an Online Learning Platform used by nurses to improve the results of a blood culture technique. The online learning tool is studied in two of four internal medicine units of a tertiary hospital in Madrid. These two units have similar characteristics of personnel, materials and structure. Both units are at a great distance, preventing a professional talk to each other.

ELIGIBILITY:
Inclusion Criteria:

* Be nurse of the nursing unit selected.
* Foreseeing to remain in service during the study.
* Acceptance of voluntary participation in the study, prior information.
* Signature of informed consent.

Exclusion Criteria:

* Those professionals who for reasons beyond their control are transferred to other services or are on leave (in any form). They can not complete the various phases of the study.
* Professionals who, for whatever reason, decide to withdraw their consent to participate in the study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Zaragoza GArcía, PhD, Principal Investigator — Hospital 12 de Octubre de Madrid
Locations (1):
- Hospital Universitario 12 de Octubre de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Not Receive Online Training: Participants don´t receives an individual online training of extraction of blood culture. Do their work as usual.
Period: Overall Study
Arm/Group | Online Training of a Nursing Technique | Not Receive Online Training
Started | 26 | 22
Completed | 26 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Nurses working in internal medicine of the "Hospital 12 de Octubre Madrid"
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Training of a Nursing Technique | Not Receive Online Training | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.08 (8.8) | 39.77 (8.03) | 39.86 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Spain | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Contaminated Cultures in the Control and Experimental Group Before Intervention and After the Learning Obtained With the Online Training Platform.
Description: The results obtained in each arm of the study are collected month by month in both groups (Experimental and control). The data for each month are summarized for 6 months, reporting the pre-intervention result (for both groups: experimental and control). The data collected during the 3 months following the intervention are also summed during the 3 months, giving a value at the end of this time (month 9 of the study).
Time Frame: assessed monthly, month 6 and 9 reported.
Population: Number of Blood culture extracted. Any blood culture is likely to be contaminated by an inadequate technique.
Measure: Number; unit: Contaminated blood cultures
Units Other Than Participants: Blood cultures
Groups:
- Online Training of a Nursing Technique Before Intervention.: Participants perform the technique of blood culture extraction in a conventional way. After 6 months of monitoring of contaminated blood cultures, this group will receive online training to improve the performance of this technique.
  Report of month 6 (amount of the first 6 months).
- Not Received Online Training Before Intervention.: Participants perform the technique of blood culture extraction in a conventional way. This group will not receives an individual online training of extraction of blood culture in any time during the study. Perform the technique as usual way.
  Report of month 6 (amount of the first 6 months).
- Online Training of a Nursing Technique After Intervention.: Participants receives an individual online training of extraction of blood culture for 3 months (This platform aims to improve knowledge and skills), they are sent 3 homework (one per month) and are evaluated at the end of each.
  Online training of a nursing technique: The professionals with participant in the experimental arm receive an online training of a technique of extraction of blood culture and other arm ("Not receive online training after intervention") They will not receive any training. They work as usual.
  Report of month 9 (amount between the 6 to 9 months).
- Not Received Online Training After Intervention.: Participants don´t receives an individual online training of extraction of blood culture.Do their work as usual.
  Report of month 9 (amount between the 6 to 9 months).
Arm/Group | Online Training of a Nursing Technique Before Intervention. | Not Received Online Training Before Intervention. | Online Training of a Nursing Technique After Intervention. | Not Received Online Training After Intervention.
Number analyzed (Participants) | 26 | 22 | 26 | 22
Number analyzed (Blood cultures) | 258 | 325 | 168 | 158
Contaminated blood cultures | 17 | 15 | 5 | 15

2. Secondary Outcome: Score on the Knowledge Test Related to Blood Culture Extraction Technique for Nurses (K-Blood-CT)
Description: The improvement in the learning of the technique is measured with a test with 20 questions created ad hoc related of blood culture intervention (Blood culture collection knowledge test for nurses). The score ranges from 0 points (worst level of knowledge) to 10 points (best level of knowledge). The results can be divided into intervals: 0-2.99 very deficient; 3- 4.99 insufficient; 5-6.9 good; 7-8.9 notable; > 9 outstanding.
Time Frame: 6 month and 9 month of study.
Population: Nurses who Work in the Internal Medicine Service of university hospital 12 de Octubre Madrid.
Measure: Mean (Standard Deviation); unit: Score on K-Blood-CT test
Groups:
- Online Training of a Nursing Technique Before Intervention.: Participants don´t receives any added knowledge or training in the 6 month before intervention. Maintain a regular training within their professional recycling. Those professionals were avaluated before starting the intervention for to know the previous level of Knowledge.
- Not Received Online Training Before Intervention.: Participants don´t receives an individual online training of extraction of blood culture.Do their work as usual. Maintain a regular training within their professional recycling. Those professionals were avaluated before starting the intervention for to know the previous level of Knowledge.
- Online Training of a Nursing Technique After Intervention.: Participants receives an individual online training of extraction of blood culture for 3 months (This platform aims to improve knowledge and skills), they are sent 3 homework (one per month) and are evaluated at the end of each.
  Online training of a nursing technique: The professionals with participant in the experimental arm receive an online training of a technique of extraction of blood culture and other arm the professionals no receive any training. They work as usual.
  Those professionals were evaluated after finished the intervention for to know the level of Knowledge.
- Not Received Online Training After Intervention.: Participants don´t receives an individual online training of extraction of blood culture.Do their work as usual.Maintain a regular training within their professional recycling.
  Those professionals were evaluated after finished the intervention for to know the level of Knowledge.
Arm/Group | Online Training of a Nursing Technique Before Intervention. | Not Received Online Training Before Intervention. | Online Training of a Nursing Technique After Intervention. | Not Received Online Training After Intervention.
Number analyzed (Participants) | 26 | 22 | 26 | 22
Score on K-Blood-CT test | 4.62 (1.57) | 4.88 (0.86) | 8.2 (0.72) | 4.6 (0.9)

ADVERSE EVENTS:
Arm/Group | Online Training of a Nursing Technique | Not Receive Online Training
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes